CLINICAL TRIAL: NCT05786729
Title: Effects of Aerobic Exercise and Rehabilitation After Traumatic Brain Injury
Brief Title: Aerobic Exercise After Traumatic Brain Injury
Acronym: AER-TBI1
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre for Neuro Skills (Industry)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Grace S. Griesbach, National Director of Clinical Research, Centre for Neuro Skills
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00016168
Record Dates: First submitted 2022-03-16; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Exercise; Rehabilitation

STUDY DESIGN:
Intervention Model Description: Intervention will consist of aerobic exercise sessions at predetermined heart rate range.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Aerobic Exercise (AER) (Experimental): Consented participants will be randomly assigned to aerobic exercise regimen (AER) + Standard Rehabilitation(R+AER) or Standard Rehabilitation only (R) group. In order to determine the necessary time window for AER exercise treatment, TBI subjects will partake in supervised AER sessions for a period of 12 weeks. After a baseline evaluations follow-ups will take place at take place at weeks 4, 8 and 12. Thus each participants will be evaluated 4 times.
  Interventions: Other: Aerobic Exercise (AER)
- Rehabilitation (R) (Active Comparator): Participants with traumatic brain injury that are enrolled in a comprehensive rehabilitation program. These participants will receive standard rehabilitation. Given that the duration of the rehabilitative program is variable the duration of participation will be no less than 4 weeks and will not exceed 12 weeks. Activity levels will be monitored.
  Interventions: Other: Rehabilitation
- Control (C) (No Intervention): Healthy volunteers' responsiveness to exercise will be compared to TBI responsiveness.

INTERVENTIONS:
Other: Aerobic Exercise (AER) — Aerobic exercise will be performed by utilizing aerobic exercise equipment 3 times per week.
  Arms: Intervention Aerobic Exercise (AER)
Other: Rehabilitation — Rehabilitative program is focused on completion of activities of daily living, initiation, appropriate behavior and community integration for five days per week at the Centre for Neuro Skills.
  Arms: Rehabilitation (R)

SUMMARY:
The purpose of this study is to examine the effects of individualized aerobic exercise regimen on recovery after traumatic brain injury (TBI).Investigators will determine if exercise facilitates recovery by facilitating neuroplasticity and decreasing neuroinflammation.

DETAILED DESCRIPTION:
Exercise-based therapies can promote recovery of function and are easily implemented in the clinical rehabilitation setting. This study will determine if exercise facilitates recovery by improving markers of neuroplasticity and decreasing neuroinflammatory responses. The investigators will also determine if variations in genes involved in neuroplasticity, and inflammation influence the responsiveness to exercise and rehabilitation. Recovery will be determined by assessing cognitive function, life quality and balance.

ELIGIBILITY:
Inclusion Criteria:

* All participants will provide informed consent and have to comply with the procedures of the study.
* Age will range from 18 to 60 years.
* Except for the non-injured control group, subjects will be required to have experienced TBI.
* All participants should be fluent in English or Spanish.
* All participants should have the ability to comply with the research protocol.
* Capable of exercising in aerobic exercise equipment (with or without trunk support).
* Able to walk independently with or without a device

Exclusion Criteria:

* Current diagnosis of degenerative neurological disease.
* A history of cerebral vascular accidents.
* A history of major psychosis as defined by DSM-IV.
* Subjects receiving physical therapy in a location that is not CNS.
* Pregnancy.
* A history of previous TBI requiring hospitalization.
* Inability to cooperate
* Orthopedic impairment that compromises exercise performance
* Any cardiovascular or respiratory condition that jeopardizes patient health during exercise.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2027-01-18 (Estimated); Study Completion 2028-01-18 (Estimated)

PRIMARY OUTCOMES:
Aerobic Exercise Induced Changes in Cardio Pulmonary Exercise (CPET) at baseline | Baseline
  CPET will allow us to determine oxygen consumption (VO2). Results will be reported as change in VO2 levels.
Aerobic Exercise Induced Changes in Cardio Pulmonary Exercise (CPET) at Week 4 | Week 4
  CPET will allow us to determine oxygen consumption (VO2). Results will be reported as change in VO2 levels.
Aerobic Exercise Induced Changes in Cardio Pulmonary Exercise (CPET) at Week 8 | Week 8
  CPET will allow us to determine oxygen consumption (VO2). Results will be reported as change in VO2 levels.
Aerobic Exercise Induced Changes in Cardio Pulmonary (CPET) at Week 12 | Week 12
  CPET will allow us to determine oxygen consumption (VO2). Results will be reported as change in VO2 levels.

SECONDARY OUTCOMES:
Aerobic Exercise Induced Changes in Cognitive Function at baseline | Baseline
  Attention, processing speed, reaction times, memory and nonverbal reasoning are evaluated by CNS Vital Signs. All scores are aggregated to one reported value (Neurocognitive Index). Scoring is by a computer based auto-scored multivariate scoring system developed by the manufacturers.
Aerobic Exercise Induced Changes in Cognitive Function at Week 4 | Week 4
  Attention, processing speed, reaction times, memory and nonverbal reasoning are evaluated by CNS Vital Signs. All scores are aggregated to one reported value (Neurocognitive Index). Scoring is by a computer based auto-scored multivariate scoring system developed by the manufacturers.
Aerobic Exercise Induced Changes in Cognitive Function at Week 8 | Week 8
  Attention, processing speed, reaction times, memory and nonverbal reasoning are evaluated by CNS Vital Signs. All scores are aggregated to one reported value (Neurocognitive Index). Scoring is by a computer based auto-scored multivariate scoring system developed by the manufacturers.
Aerobic Exercise Induced Changes in Cognitive Function at Week 12 | Week 12
  Attention, processing speed, reaction times, memory and nonverbal reasoning are evaluated by CNS Vital Signs. All scores are aggregated to one reported value (Neurocognitive Index). Scoring is by a computer based auto-scored multivariate scoring system developed by the manufacturers.
Verbal Memory Assessed by the California Verbal Learning Test (CVLT II) at baseline | Baseline
  The California Verbal Learning Test (CVLT II) is a verbal memory cognitive assessment. It assesses repetition learning, serial position effects, semantic organization, intrusions, and proactive interference. CVLT II scores have a mean of 0 and a SD of 1. The range of scores is +5 to -5 reported in increments of .5.
Verbal Memory Assessed by the California Verbal Learning Test (CVLT II) at Week 4 | Week 4
  The California Verbal Learning Test (CVLT II) is a verbal memory cognitive assessment. It assesses repetition learning, serial position effects, semantic organization, intrusions, and proactive interference. CVLT II scores have a mean of 0 and a SD of 1. The range of scores is +5 to -5 reported in increments of .5.
Verbal Memory Assessed by the California Verbal Learning Test (CVLT II) at Week 8 | Week 8
  The California Verbal Learning Test (CVLT II) is a verbal memory cognitive assessment. It assesses repetition learning, serial position effects, semantic organization, intrusions, and proactive interference. CVLT II scores have a mean of 0 and a SD of 1. The range of scores is +5 to -5 reported in increments of .5.
Verbal Memory Assessed by the California Verbal Learning Test (CVLT II) at Week 12 | Week 12
  The California Verbal Learning Test (CVLT II) is a verbal memory cognitive assessment. It assesses repetition learning, serial position effects, semantic organization, intrusions, and proactive interference. CVLT II scores have a mean of 0 and a SD of 1. The range of scores is +5 to -5 reported in increments of .5.
Quality of Life Measured by the NeuroQOL at baseline | Baseline
  The NeuroQOL assesses quality of life in the domains of Physical Domain, Mental Domain, Cognitive Domain, and Social Domain. Items are scored on a 5-point scale that uses different language depending on assessment. The questions range from least (1) to most (5) based on frequency of behavior, amount of difficulty, or degree of agreement. T-score are used, mean of 50 and SD of 10
Quality of Life Measured by the NeuroQOL at Week 4 | Week 4
  The NeuroQOL assesses quality of life in the domains of Physical Domain, Mental Domain, Cognitive Domain, and Social Domain. Items are scored on a 5-point scale that uses different language depending on assessment. The questions range from least (1) to most (5) based on frequency of behavior, amount of difficulty, or degree of agreement. T-score are used, mean of 50 and SD of 10
Quality of Life Measured by the NeuroQOL at Week 8 | Week 8
  The NeuroQOL assesses quality of life in the domains of Physical Domain, Mental Domain, Cognitive Domain, and Social Domain. Items are scored on a 5-point scale that uses different language depending on assessment. The questions range from least (1) to most (5) based on frequency of behavior, amount of difficulty, or degree of agreement. T-score are used, mean of 50 and SD of 10
Quality of Life Measured by the NeuroQOL at Week 12 | Week 12
  The NeuroQOL assesses quality of life in the domains of Physical Domain, Mental Domain, Cognitive Domain, and Social Domain. Items are scored on a 5-point scale that uses different language depending on assessment. The questions range from least (1) to most (5) based on frequency of behavior, amount of difficulty, or degree of agreement. T-score are used, mean of 50 and SD of 10
Depression measured by the Beck Depression Inventory-II at baseline | Baseline
  The Beck Depression Inventory- II (BDI-II) assesses depressive symptom severity. The BDI-II is comprised of 21 individual items reflecting specific cognitive, affective, and physical symptoms of depression. Each item includes four statements that vary in the description of symptom of severity. Scores range from 0 to 3, with a score of "3" indicating a severe symptoms and a score of "0" indicating an absence of concern with that particular aspect of depressive symptomology. The total score is the sum of all endorsed statements. The maximum total score is 63. The BDI-II Manual designates the following raw score classifications depression severity: ≤13 = minimal; 14-19 = mild; 20-28 = moderate; ≥ 29 = severe.
Depression measured by the Beck Depression Inventory-II at Week 4 | Week 4
  The Beck Depression Inventory- II (BDI-II) assesses depressive symptom severity. The BDI-II is comprised of 21 individual items reflecting specific cognitive, affective, and physical symptoms of depression. Each item includes four statements that vary in the description of symptom of severity. Scores range from 0 to 3, with a score of "3" indicating a severe symptoms and a score of "0" indicating an absence of concern with that particular aspect of depressive symptomology. The total score is the sum of all endorsed statements. The maximum total score is 63. The BDI-II Manual designates the following raw score classifications depression severity: ≤13 = minimal; 14-19 = mild; 20-28 = moderate; ≥ 29 = severe.
Depression measured by the Beck Depression Inventory-II at Week 8 | Week 8
  The Beck Depression Inventory- II (BDI-II) assesses depressive symptom severity. The BDI-II is comprised of 21 individual items reflecting specific cognitive, affective, and physical symptoms of depression. Each item includes four statements that vary in the description of symptom of severity. Scores range from 0 to 3, with a score of "3" indicating a severe symptoms and a score of "0" indicating an absence of concern with that particular aspect of depressive symptomology. The total score is the sum of all endorsed statements. The maximum total score is 63. The BDI-II Manual designates the following raw score classifications depression severity: ≤13 = minimal; 14-19 = mild; 20-28 = moderate; ≥ 29 = severe.
Depression measured by the Beck Depression Inventory-II at Week 12 | Week 12
  The Beck Depression Inventory- II (BDI-II) assesses depressive symptom severity. The BDI-II is comprised of 21 individual items reflecting specific cognitive, affective, and physical symptoms of depression. Each item includes four statements that vary in the description of symptom of severity. Scores range from 0 to 3, with a score of "3" indicating a severe symptoms and a score of "0" indicating an absence of concern with that particular aspect of depressive symptomology. The total score is the sum of all endorsed statements. The maximum total score is 63. The BDI-II Manual designates the following raw score classifications depression severity: ≤13 = minimal; 14-19 = mild; 20-28 = moderate; ≥ 29 = severe.
Visual Search/ Processing Speed measured by Trail Making Test (TMT) at baseline | Baseline
  The Trail Making Test (TMT) provides information on visual search, scanning, speed of processing, mental flexibility, and executive functions. The TMT consists of two parts. TMT-A requires an individual to draw lines sequentially connecting 25 encircled numbers distributed on a sheet of paper. Task requirements are similar for TMT-B except the person must alternate between numbers and letters (e.g., 1, A, 2, B, 3, C, etc.). The score on each part represents the amount of time required to complete the task.
Visual Search/ Processing Speed measured by Trail Making Test (TMT) at Week 4 | Week 4
  The Trail Making Test (TMT) provides information on visual search, scanning, speed of processing, mental flexibility, and executive functions. The TMT consists of two parts. TMT-A requires an individual to draw lines sequentially connecting 25 encircled numbers distributed on a sheet of paper. Task requirements are similar for TMT-B except the person must alternate between numbers and letters (e.g., 1, A, 2, B, 3, C, etc.). The score on each part represents the amount of time required to complete the task.
Visual Search/ Processing Speed measured by Trail Making Test (TMT) at Week 8 | Week 8
  The Trail Making Test (TMT) provides information on visual search, scanning, speed of processing, mental flexibility, and executive functions. The TMT consists of two parts. TMT-A requires an individual to draw lines sequentially connecting 25 encircled numbers distributed on a sheet of paper. Task requirements are similar for TMT-B except the person must alternate between numbers and letters (e.g., 1, A, 2, B, 3, C, etc.). The score on each part represents the amount of time required to complete the task.
Visual Search/ Processing Speed measured by Trail Making Test (TMT) at Week 12 | Week 12
  The Trail Making Test (TMT) provides information on visual search, scanning, speed of processing, mental flexibility, and executive functions. The TMT consists of two parts. TMT-A requires an individual to draw lines sequentially connecting 25 encircled numbers distributed on a sheet of paper. Task requirements are similar for TMT-B except the person must alternate between numbers and letters (e.g., 1, A, 2, B, 3, C, etc.). The score on each part represents the amount of time required to complete the task.
Sleepiness will be measured by the Epworth Sleepiness Scale at baseline | Baseline
  The Epworth Sleepiness Scale is used to measure a patient's sleepiness. The test is a list of eight situations in which the patient rates their tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing. Total score is based on a scale of 0 to 24. The scale estimates whether you are experiencing excessive sleepiness.
Sleepiness will be measured by the Epworth Sleepiness Scale at Week 4 | Week 4
  The Epworth Sleepiness Scale is used to measure a patient's sleepiness. The test is a list of eight situations in which the patient rates their tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing. Total score is based on a scale of 0 to 24. The scale estimates whether you are experiencing excessive sleepiness.
Sleepiness will be measured by the Epworth Sleepiness Scale at Week 8 | Week 8
  The Epworth Sleepiness Scale is used to measure a patient's sleepiness. The test is a list of eight situations in which the patient rates their tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing. Total score is based on a scale of 0 to 24. The scale estimates whether you are experiencing excessive sleepiness.
Sleepiness will be measured by the Epworth Sleepiness Scale at Week 12 | Week 12
  The Epworth Sleepiness Scale is used to measure a patient's sleepiness. The test is a list of eight situations in which the patient rates their tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing. Total score is based on a scale of 0 to 24. The scale estimates whether you are experiencing excessive sleepiness.
Vestibular function will be measured by the Berg Balance Test at baseline | Baseline
  The Berg Balance Scale is used to determine vestibular function through a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function.
Vestibular function will be measured by the Berg Balance Test at Week 4 | Week 4
  The Berg Balance Scale is used to determine vestibular function through a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function.
Vestibular function will be measured by the Berg Balance Test at Week 8 | Week 8
  The Berg Balance Scale is used to determine vestibular function through a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function.
Vestibular function will be measured by the Berg Balance Test at Week 12 | Week 12
  The Berg Balance Scale is used to determine vestibular function through a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function.
Aerobic capacity and endurance will be measured with the 6 Minute Walk Test at baseline | Baseline
  The 6 Minute Walk Test (6MWT) is a exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway. A lower score (reflecting less distance covered in 6 minutes) indicates worse function. An increase in the distance walked indicates improvement in basic mobility.
Aerobic capacity and endurance will be measured with the 6 Minute Walk Test at Week 4 | Week 4
  The 6 Minute Walk Test (6MWT) is a exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway. A lower score (reflecting less distance covered in 6 minutes) indicates worse function. An increase in the distance walked indicates improvement in basic mobility.
Aerobic capacity and endurance will be measured with the 6 Minute Walk Test at Week 8 | Week 8
  The 6 Minute Walk Test (6MWT) is a exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway. A lower score (reflecting less distance covered in 6 minutes) indicates worse function. An increase in the distance walked indicates improvement in basic mobility.
Aerobic capacity and endurance will be measured with the 6 Minute Walk Test at Week 12 | Week 12
  The 6 Minute Walk Test (6MWT) is a exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway. A lower score (reflecting less distance covered in 6 minutes) indicates worse function. An increase in the distance walked indicates improvement in basic mobility.
Evaluation of Inflammatory Biomarkers at Baseline | Baseline
  Biomarkers IL10, IL12, IL-1β, IL-4 , IL-5, IL-6, IL-7, IL-8, TNFα, will be measured in blood serum before and after a 30 minute aerobic activity. Results will be reported as change in levels.
Evaluation of Inflammatory Biomarkers at Week 4 | Week 4
  Biomarkers IL10, IL12, IL-1β, IL-4 , IL-5, IL-6, IL-7, IL-8, TNFα, will be measured in blood serum before and after a 30 minute aerobic activity. Results will be reported as change in levels.
Evaluation of Inflammatory Biomarkers at Week 8 | Week 8
  Biomarkers IL10, IL12, IL-1β, IL-4 , IL-5, IL-6, IL-7, IL-8, TNFα, will be measured in blood serum before and after a 30 minute aerobic activity. Results will be reported as change in levels.
Evaluation of Inflammatory Biomarkers at Week 12 | Week 12
  Biomarkers IL10, IL12, IL-1β, IL-4 , IL-5, IL-6, IL-7, IL-8, TNFα, will be measured in blood serum before and after a 30 minute aerobic activity. Results will be reported as change in levels.
Evaluation of Neuroplasticity, Stress Biomarkers at Baseline | Baseline
  Biomarkers BDNF, GH, ACTH, Cortisol, Melatonin, VEGF will be measured in blood serum before and after a 30 minute aerobic activity. Results will be reported as change in levels.
Evaluation of Neuroplasticity, Stress Biomarkers at Week 4 | Week 4
  Biomarkers BDNF, GH, ACTH, Cortisol, Melatonin, VEGF will be measured in blood serum before and after a 30 minute aerobic activity. Results will be reported as change in levels.
Evaluation of Neuroplasticity, Stress Biomarkers at Week 8 | Week 8
  Biomarkers BDNF, GH, ACTH, Cortisol, Melatonin, VEGF will be measured in blood serum before and after a 30 minute aerobic activity. Results will be reported as change in levels.
Evaluation of Neuroplasticity, Stress Biomarkers at Week 12 | Week 12
  Biomarkers BDNF, GH, ACTH, Cortisol, Melatonin, VEGF will be measured in blood serum before and after a 30 minute aerobic activity. Results will be reported as change in levels.
Evaluation of Neurodegeneration Biomarkers at Baseline | Baseline
  Biomarkers sCAM1, vCAM-1, sFAS will be measured in blood serum before and after a 30 minute aerobic activity. Results will be reported as change in levels.
Evaluation of Neurodegeneration Biomarkers at Week 4 | Week 4
  Biomarkers sCAM1, vCAM-1, sFAS will be measured in blood serum before and after a 30 minute aerobic activity. Results will be reported as change in levels.
Evaluation of Neurodegeneration Biomarkers at Week 8 | Week 8
  Biomarkers sCAM1, vCAM-1, sFAS will be measured in blood serum before and after a 30 minute aerobic activity. Results will be reported as change in levels.
Evaluation of Neurodegeneration Biomarkers at Week 12 | Week 12
  Biomarkers sCAM1, vCAM-1, sFAS will be measured in blood serum before and after a 30 minute aerobic activity. Results will be reported as change in levels.
BDNF / Val66Met at baseline | Baseline
  Evaluation of genetic material BDNF / Val66Met will be measured in a saliva sample. Results will be reported as% difference from the general population.
BDNF / Val66Met at Week 4 | Week 4
  Evaluation of genetic material BDNF / Val66Met will be measured in a saliva sample. Results will be reported as% difference from the general population.
BDNF / Val66Met at Week 8 | Week 8
  Evaluation of genetic material BDNF / Val66Met will be measured in a saliva sample. Results will be reported as% difference from the general population.
BDNF / Val66Met at Week 12 | Week 12
  Evaluation of genetic material BDNF / Val66Met will be measured in a saliva sample. Results will be reported as% difference from the general population.
IL-1β / rs16944 at baseline | Baseline
  Evaluation of genetic material IL-1β / rs16944 will be measured in a saliva sample. Results will be reported as% difference from the general population.
IL-1β / rs16944 at Week 4 | Week 4
  Evaluation of genetic material IL-1β / rs16944 will be measured in a saliva sample. Results will be reported as% difference from the general population.
IL-1β / rs16944 at Week 8 | Week 8
  Evaluation of genetic material IL-1β / rs16944 will be measured in a saliva sample. Results will be reported as% difference from the general population.
IL-1β / rs16944 at Week 12 | Week 12
  Evaluation of genetic material IL-1β / rs16944 will be measured in a saliva sample. Results will be reported as% difference from the general population.
TrkB at baseline | Baseline
  Evaluation of genetic material TrkB will be measured in a saliva sample. Results will be reported as% difference from the general population.
TrkB at Week 4 | Week 4
  Evaluation of genetic material TrkB will be measured in a saliva sample. Results will be reported as% difference from the general population.
TrkB at Week 8 | Week 8
  Evaluation of genetic material TrkB will be measured in a saliva sample. Results will be reported as% difference from the general population.
TrkB at Week 12 | Week 12
  Evaluation of genetic material TrkB will be measured in a saliva sample. Results will be reported as% difference from the general population.
COMT / VAll58Met at baseline | Baseline
  Evaluation of genetic material COMT / VAll58Met will be measured in a saliva sample. Results will be reported as% difference from the general population.
COMT / VAll58Met at Week 4 | Week 4
  Evaluation of genetic material COMT / VAll58Met will be measured in a saliva sample. Results will be reported as% difference from the general population.
COMT / VAll58Met at Week 8 | Week 8
  Evaluation of genetic material COMT / VAll58Met will be measured in a saliva sample. Results will be reported as% difference from the general population.
COMT / VAll58Met at Week 12 | Week 12
  Evaluation of genetic material COMT / VAll58Met ewill be measured in a saliva sample. Results will be reported as% difference from the general population.
DRD2 / A to T & A to G at baseline | Baseline
  Evaluation of genetic material DRD2 / A to T & A to G will be measured in a saliva sample. Results will be reported as% difference from the general population.
DRD2 / A to T & A to G at Week 4 | Week 4
  Evaluation of genetic material DRD2 / A to T & A to G will be measured in a saliva sample. Results will be reported as% difference from the general population.
DRD2 / A to T & A to G at Week 8 | Week 8
  Evaluation of genetic material DRD2 / A to T & A to G will be measured in a saliva sample. Results will be reported as% difference from the general population.
DRD2 / A to T & A to G at Week 12 | Week 12
  Evaluation of genetic material DRD2 / A to T & A to G will be measured in a saliva sample. Results will be reported as% difference from the general population.
ANKKI / TAQIA at baseline | Baseline
  Evaluation of genetic material ANKKI / TAQIA will be measured in a saliva sample. Results will be reported as% difference from the general population.
ANKKI / TAQIA at Week 4 | Week 4
  Evaluation of genetic material ANKKI / TAQIA will be measured in a saliva sample. Results will be reported as% difference from the general population.
ANKKI / TAQIA at Week 8 | Week 8
  Evaluation of genetic material ANKKI / TAQIA will be measured in a saliva sample. Results will be reported as% difference from the general population.
ANKKI / TAQIA at Week 12 | Week 12
  Evaluation of genetic material ANKKI / TAQIA will be measured in a saliva sample. Results will be reported as% difference from the general population.
PPPIRIB / C to T at baseline | Baseline
  Evaluation of genetic material PPPIRIB / C to T will be measured in a saliva sample. Results will be reported as% difference from the general population.
PPPIRIB / C to T at Week 4 | week 4
  Evaluation of genetic material PPPIRIB / C to T will be measured in a saliva sample. Results will be reported as% difference from the general population.
PPPIRIB / C to T at Week 8 | week 8
  Evaluation of genetic material PPPIRIB / C to T will be measured in a saliva sample. Results will be reported as% difference from the general population.
PPPIRIB / C to T at Week 12 | week 12
  Evaluation of genetic material PPPIRIB / C to T will be measured in a saliva sample. Results will be reported as% difference from the general population.
MAO-A /MAOA-H & MAOA-L at baseline | Baseline
  Evaluation of genetic material MAO-A /MAOA-H & MAOA-L will be measured in a saliva sample. Results will be reported as% difference from the general population.
MAO-A /MAOA-H & MAOA-L at Week 4 | Week 4
  Evaluation of genetic material MAO-A /MAOA-H & MAOA-L will be measured in a saliva sample. Results will be reported as% difference from the general population.
MAO-A /MAOA-H & MAOA-L at Week 8 | Week 8
  Evaluation of genetic material MAO-A /MAOA-H & MAOA-Lwill be measured in a saliva sample. Results will be reported as% difference from the general population.
MAO-A /MAOA-H & MAOA-L at Week 12 | Week 12
  Evaluation of genetic material MAO-A /MAOA-H & MAOA-L will be measured in a saliva sample. Results will be reported as% difference from the general population.
5-HTR2A / AI438G at baseline | Baseline
  Evaluation of genetic material 5-HTR2A / AI438G will be measured in a saliva sample. Results will be reported as % difference from the general population.
5-HTR2A / AI438G at Week 4 | Week 4
  Evaluation of genetic material 5-HTR2A / AI438G will be measured in a saliva sample. Results will be reported as% difference from the general population.
5-HTR2A / AI438G at Week 8 | Week 8
  Evaluation of genetic material 5-HTR2A / AI438G will be measured in a saliva sample. Results will be reported as% difference from the general population.
5-HTR2A / AI438G at Week 12 | Week 12
  Evaluation of genetic material 5-HTR2A / AI438G will be measured in a saliva sample. Results will be reported as% difference from the general population.
5-HT1A / C1019G at baseline | Baseline
  Evaluation of genetic material 5-HT1A / C1019G will be measured in a saliva sample. Results will be reported as% difference from the general population.
5-HT1A / C1019G at Week 4 | Week 4
  Evaluation of genetic material 5-HT1A / C1019G will be measured in a saliva sample. Results will be reported as% difference from the general population.
5-HT1A / C1019G at Week 8 | Week 8
  Evaluation of genetic material 5-HT1A / C1019G will be measured in a saliva sample. Results will be reported as% difference from the general population.
5-HT1A / C1019G at Week 12 | Week 12
  Evaluation of genetic material 5-HT1A / C1019G will be measured in a saliva sample. Results will be reported as% difference from the general population.
5-HTR2B / HTR2B Q20 at baseline | Baseline
  Evaluation of genetic material 5-HTR2B / HTR2B Q20 will be measured in a saliva sample. Results will be reported as% difference from the general population.
5-HTR2B / HTR2B Q20 at Week 4 | Week 4
  Evaluation of genetic material 5-HTR2B / HTR2B Q20 will be measured in a saliva sample. Results will be reported as% difference from the general population.
5-HTR2B / HTR2B Q20 at Week 8 | Week 8
  Evaluation of genetic material 5-HTR2B / HTR2B Q20 will be measured in a saliva sample. Results will be reported as% difference from the general population.
5-HTR2B / HTR2B Q20 at Week 12 | Week 12
  Evaluation of genetic material 5-HTR2B / HTR2B Q20 will be measured in a saliva sample. Results will be reported as% difference from the general population.
TPH / A218C & A779C at baseline | Baseline
  Evaluation of genetic material TPH / A218C & A779C will be measured in a saliva sample. Results will be reported as% difference from the general population.
TPH / A218C & A779C at Week 4 | Week 4
  Evaluation of genetic material TPH / A218C & A779C will be measured in a saliva sample. Results will be reported as% difference from the general population.
TPH / A218C & A779C at Week 8 | Week 8
  Evaluation of genetic material TPH / A218C & A779C will be measured in a saliva sample. Results will be reported as% difference from the general population.
TPH / A218C & A779C at Week 12 | Week 12
  Evaluation of genetic material TPH / A218C & A779C will be measured in a saliva sample. Results will be reported as% difference from the general population.

CONTACTS AND LOCATIONS:
Overall Officials: Grace S Griesbach, PhD, Principal Investigator — Centre for Neuro Skills
Locations (1):
- Centre for Neuro Skills, Bakersfield, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ashman TA, Gordon WA, Cantor JB, Hibbard MR. Neurobehavioral consequences of traumatic brain injury. Mt Sinai J Med. 2006 Nov;73(7):999-1005. PMID 17195886
- [Background] Kleim JA, Jones TA, Schallert T. Motor enrichment and the induction of plasticity before or after brain injury. Neurochem Res. 2003 Nov;28(11):1757-69. doi: 10.1023/a:1026025408742. PMID 14584829
- [Background] Griesbach GS, Hovda DA, Molteni R, Wu A, Gomez-Pinilla F. Voluntary exercise following traumatic brain injury: brain-derived neurotrophic factor upregulation and recovery of function. Neuroscience. 2004;125(1):129-39. doi: 10.1016/j.neuroscience.2004.01.030. PMID 15051152
- [Background] Griesbach GS, Hovda DA, Gomez-Pinilla F. Exercise-induced improvement in cognitive performance after traumatic brain injury in rats is dependent on BDNF activation. Brain Res. 2009 Sep 8;1288:105-15. doi: 10.1016/j.brainres.2009.06.045. Epub 2009 Jun 23. PMID 19555673
- [Background] Seifert T, Brassard P, Wissenberg M, Rasmussen P, Nordby P, Stallknecht B, Adser H, Jakobsen AH, Pilegaard H, Nielsen HB, Secher NH. Endurance training enhances BDNF release from the human brain. Am J Physiol Regul Integr Comp Physiol. 2010 Feb;298(2):R372-7. doi: 10.1152/ajpregu.00525.2009. Epub 2009 Nov 18. PMID 19923361
- [Background] Johnson VE, Stewart W, Smith DH. Axonal pathology in traumatic brain injury. Exp Neurol. 2013 Aug;246:35-43. doi: 10.1016/j.expneurol.2012.01.013. Epub 2012 Jan 20. PMID 22285252
- [Background] Povlishock JT, Pettus EH. Traumatically induced axonal damage: evidence for enduring changes in axolemmal permeability with associated cytoskeletal change. Acta Neurochir Suppl. 1996;66:81-6. doi: 10.1007/978-3-7091-9465-2_15. PMID 8780803
- [Background] Schuit AJ, Feskens EJ, Launer LJ, Kromhout D. Physical activity and cognitive decline, the role of the apolipoprotein e4 allele. Med Sci Sports Exerc. 2001 May;33(5):772-7. doi: 10.1097/00005768-200105000-00015. PMID 11323547
- [Background] Adlard PA, Perreau VM, Pop V, Cotman CW. Voluntary exercise decreases amyloid load in a transgenic model of Alzheimer's disease. J Neurosci. 2005 Apr 27;25(17):4217-21. doi: 10.1523/JNEUROSCI.0496-05.2005. PMID 15858047
- [Background] Piao CS, Stoica BA, Wu J, Sabirzhanov B, Zhao Z, Cabatbat R, Loane DJ, Faden AI. Late exercise reduces neuroinflammation and cognitive dysfunction after traumatic brain injury. Neurobiol Dis. 2013 Jun;54:252-63. doi: 10.1016/j.nbd.2012.12.017. Epub 2013 Jan 8. PMID 23313314
- [Background] Norden DM, Muccigrosso MM, Godbout JP. Microglial priming and enhanced reactivity to secondary insult in aging, and traumatic CNS injury, and neurodegenerative disease. Neuropharmacology. 2015 Sep;96(Pt A):29-41. doi: 10.1016/j.neuropharm.2014.10.028. Epub 2014 Nov 13. PMID 25445485
- [Background] Gurley JM, Hujsak BD, Kelly JL. Vestibular rehabilitation following mild traumatic brain injury. NeuroRehabilitation. 2013;32(3):519-28. doi: 10.3233/NRE-130874. PMID 23648606
- [Background] Rinne MB, Pasanen ME, Vartiainen MV, Lehto TM, Sarajuuri JM, Alaranta HT. Motor performance in physically well-recovered men with traumatic brain injury. J Rehabil Med. 2006 Jul;38(4):224-9. doi: 10.1080/16501970600582989. PMID 16801204
- [Background] Bland DC, Zampieri C, Damiano DL. Effectiveness of physical therapy for improving gait and balance in individuals with traumatic brain injury: a systematic review. Brain Inj. 2011;25(7-8):664-79. doi: 10.3109/02699052.2011.576306. Epub 2011 May 11. PMID 21561297